CLINICAL TRIAL: NCT04473781
Title: Prospective Study of Interstitial Brachytherapy for Unresectable/Unablatable T1b/T2a Renal Masses
Brief Title: Interstitial Brachytherapy for the Treatment of Unresectable/Unablatable Kidney Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-001258; NCI-2020-04542 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Stage I Renal Cell Cancer; Stage II Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (interstitial brachytherapy) (Experimental): Patients undergo interstitial brachytherapy for 1-2 fractions in the absence of disease progression or unacceptable toxicity. Patients who undergo 2 fractions may receive both fractions in the same day or on 2 separate days over 2 weeks.
  Interventions: Procedure: Interstitial Radiation Therapy

INTERVENTIONS:
Procedure: Interstitial Radiation Therapy — Undergo interstitial brachytherapy
  Other Names: BRACHYTHERAPY, INTERSTITIAL; Implant Radiation

SUMMARY:
This phase I/II trial investigates the side effects of interstitial brachytherapy and to see how well it works in limiting the growth of large kidney cancer masses in patients with kidney cancer that have refused or are unable to undergo surgery or ablation (unresectable/unablatable). Brachytherapy, also known as internal radiation therapy, temporarily introduces a radiation source into or near the tumor to eradicate the tumor cells. Giving brachytherapy may potentially reduce the size of the kidney cancer mass that would otherwise not be amenable to surgical management and translate into lower risk of spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of renal interstitial radiation therapy (interstitial brachytherapy). (Safety Lead-In) II. To evaluate local control of renal interstitial brachytherapy. (Expansion Phase)

SECONDARY OBJECTIVES:

I. To evaluate treatment response of the primary tumor. II. To evaluate 12 month distant progression free survival. III. To evaluate the 12 month volumetric growth of the primary tumor mass. IV. To determine biomarkers predicting response and resistance to radiation treatment.

OUTLINE:

Patients undergo interstitial brachytherapy for 1-2 fractions in the absence of disease progression or unacceptable toxicity. Patients who undergo 2 fractions may receive both fractions in the same day or on 2 separate days over 2 weeks.

After completion of study treatment, patients are followed up every 3 months for at least 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Elected to undergo interstitial brachytherapy as part of conventional treatment for renal cell carcinoma
* Biopsy proven renal cell carcinoma
* No definitive evidence of locally advanced (nodal or tumor thrombus) or distant (metastatic) disease
* Lesion size (maximal dimension) of 4 to 10 cm
* Patient not a candidate for curative surgery (unwilling or unable to pursue surgery)
* Lesion cannot be reliably treated with ablative techniques
* Entire lesion able to be treated adequately by brachytherapy per radiation oncologist
* Tumor predominantly solid (~ > 80%)
* Lesion that has been observed for >= 6 months with demonstrable growth rate anticipated to be >= 4 mm/year by same imaging modality
* Renal tumor that is amenable to percutaneous access for interstitial renal brachytherapy (Institutional Review Board [IRB])
* Hemoglobin > 9
* Absolute neutrophil count (ANC) >= 1500/uL (microliter)
* Platelets >= 100,000/uL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 upper limit of normal (ULN)
* Total bilirubin =< ULN
* A competent immune system
* Estimated glomerular filtration rate (eGFR) >= 30
* Good performance status (Eastern Cooperative Oncology Group [ECOG]) < 2
* Understanding and willingness to provide consent
* No prior systemic treatment for kidney cancer
* Women of childbearing potential must have negative pregnancy test at start of therapy

Exclusion Criteria:

* Presence of an active, untreated, non-renal malignancy
* Uncontrolled medical illness including infections, hypertension, arrhythmias, heart failure, or myocardial infarction within 6 months
* History of bleeding diathesis or recent bleeding episode
* Need for urgent treatment of renal cancer due bleeding, pain, or paraneoplastic syndrome
* Prior surgery or radiation therapy to the operative site
* Unwillingness to undergo clinical and laboratory monitoring and/or imaging studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | From the first administration of study therapy up to 60 days
  A 3+3 safety lead-in phase will be employed in order to determine the DLT for interstitial renal brachytherapy. Grading of DLTs will follow the guidelines provided in the Common Terminology Criteria for Adverse Events version 5.0 criteria.
One year (12-month) linear growth rate | At 1 year
  Adequate local control will be defined as minimal growth kinetics (=< 1 mm/year) on 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Chang, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States